CLINICAL TRIAL: NCT05954624
Title: A Open-Label, Two-sequence Phase I Drug-drug Interaction Clinical Study to Investigate the Pharmacokinetics of ZSP1273 With Digoxin, Rosuvastatin,Itraconazole and Probenecid in Healthy Participants
Brief Title: Drug-durg Interaction of ZSP1273 With Digoxin, Rosuvastatin,Itraconazole and Probenecid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-23-13
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium; ZSP1273; Itraconazole; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): All participants will receive the following oral doses of study drugs following an overnight fast in the fixed-sequence below:
  Period 1: 1 × 0.25-mg digoxin tablet, 1 × 10-mg rosuvastatin tablet Period 2: 8 × 600-mg ZSP1273 tablet+1 × 0.25 mg digoxin tablet, 1 × 10-mg rosuvastatin tablet
  Interventions: Drug: Digoxin; Drug: Rosuvastatin; Drug: ZSP1273
- Experimental 2 (Experimental): All participants will receive the following oral doses of study drugs following an overnight fast in the fixed-sequence below:
  Period 1: 600-mg ZSP1273 tablet Period 2: 5× 500mg Probenecid tablet BID+600-mg ZSP1273 tablet Period3: （Day1）200mg Itraconazole Capsule BID，（Day2-7）200mg Itraconazole Capsule QD+600-mg ZSP1273 tablet
  Interventions: Drug: ZSP1273; Drug: Itraconazole; Drug: Probenecid

INTERVENTIONS:
Drug: Digoxin — oral
  Arms: Experimental 1
Drug: Rosuvastatin — oral
  Arms: Experimental 1
Drug: ZSP1273 — oral
Drug: Itraconazole — oral
  Arms: Experimental 2
Drug: Probenecid — oral
  Arms: Experimental 2

SUMMARY:
The drug-drug interaction study had been designed to investigate the effect of ZSP1273 on the pharmacokinetics of digoxin, Rosuvastatin and the effect of Itraconazole and Probenecid on the pharmacokinetics of ZSP1273

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥19 to ≤26kg/m2 and total body weight >50 kg(male) or >45kg(female) at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;
3. Normal physical examination, vital signs, 12-lead ECG, and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with a history of hypersensitivity to study drug(ZSP1273,Digoxin, Rosuvastatin,Itraconazole ) or any component of study medication;
2. Participants had taken prescription, over-the-counter, herbal, or vitamin products within 28 days prior to screening；
3. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (> 400 mL) 3 months prior to randomization;
5. Those with clinically significant Electrocardiogram(ECG) abnormalities, or QTcF > 450ms;
6. Participants who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or Syphilis spirochete-specific antibodies (TPPA);
7. Participants who test positive at Screening and/or admission (Day -1) for alcohol abuse.
8. Females who are pregnant, lactating, or likely to become pregnant during the study.
9. History of dysphagia or any gastrointestinal disorder that affect absorption

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic - Cmax | 0-168 hours
  Maximum observed plasma concentration
Pharmacokinetic -Area under the curve（AUC） | 0-168 hours
  Area under the curve

SECONDARY OUTCOMES:
Number of participants with adverse events | Day1 to Day30
  The safety and tolerability of ZSP1273 alone and in combination with Itraconazole, rosuvastatin, Probenecid and digoxin will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou University of Chinese medicine, Guangzhou, China